CLINICAL TRIAL: NCT03146208
Title: Biomarkers of Coronary Artery Diseases
Brief Title: Role of Endothelial Biomarkers in Patients With Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naglaa Kamal Idriss, Doctor, Assiut University
Other Study IDs: 17200057
Record Dates: First submitted 2017-05-06; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus; Cytomegalovirus Infections
Keywords: Growth differentiation factor-15; Dipeptidyl-peptidase inhibitors (DPP4 -I); Coronroy artery diseases
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 11 Months
Biospecimen Retention: Samples With DNA — Quantitative Analysis of telomere length & GDF-15 by Real-time PCR in plasma, HUVCES, and Cell line.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Coronary artery disease patients with type 2 DM: Coronary artery disease patients with type 2 diabetes (age 20-55 years). The present study will be carried on 25 patients attending to cardiology department with coronary artery disease with type 2 diabetes
- Coronary artery disease patients without type 2 DM: The present study will be carried on 29 patients attending to cardiology department with coronary artery disease without type 2 diabetes (age 20-55 years).
- Healthy control group: we will include 54 age-matched patients with normal angiogram

SUMMARY:
Coronary artery disease is a contraction of the coronary arteries that prevent adequate blood supply to the heart muscle is called CAD. Usually caused by atherosclerosis, it may be advanced to the point where the heart muscle is injured due to lack of blood supply. Such damage may result in infarction, arrhythmias, and heart failure(1,2).

Telomeres are short in circulating leucocytes in patients with coronary artery disease but the precise mechanism is not well-known (3).

Telomere and telomerase are affected by cytomegalovirus (CMV) infection due to its effect on increasing the number of highly differentiated T cells that are characterized by shorter telomere length (TL) and lowered telomerase activity (TA). Both genetic and environmental factors have been connected with individual distinction in TL.Cardiovascular risk factors such as smoking, diabetes mellitus, hypertension, obesity, and stress have been considered to upsurge inflammation, oxidative stress, therefore accelerating TL shortening (1,2)

It has also been observed that telomere loss in type 2 diabetic patients contributes to oxidative stress and endoplasmic reticulum stress while telomere shortening has also been proposed that it can serve as an independent risk factor of T2DM and it can measure disease progression(4).

Moreover, telomeric length in peripheral blood mononuclear cells (PBMCs) is associated with the duration of disease and good glycemic control seems to be protective for telomeric loss (5).

Growth differentiation factor-15 (GDF-15) is a member of the transforming growth factor (TGF)-β superfamily. GDF-15, recently identified as one of the new cardioprotective cytokines. It is highly expressed in cardiomyocytes, adipocytes, macrophages, endothelial cells, and vascular smooth muscle cells in normal and pathological condition. GDF-15 increases during tissue injury and inflammatory states and is associated with cardiometabolic risk(6).

Dipeptidyl peptidase inhibitors (DPP4 -I) are called gliptins which increase the incretin levels and therefore prolong the post-prandial insulin action(7).

Diana et al reported that In type 2 diabetic patients, leukocyte telomere was significantly shorter than control groups and was significantly elongated after intervention by sitagliptin(8).

The common feature of all risk factors of CAD and T2DM imbalance between pro- and anti-oxidative factors in the organism with an increased production of reactive oxygen species (ROS).Nuclear factor erythroid-derived factor 2-related factor 2(Nrf2) is a family of transcription factors which plays an important role in protection against CVD and DM by regulating antioxidant enzymes in cells after ROS exposure (9).

In our study, we will propose a model, which would provide the basis to establish a marker for chronic reactivation of CMV and shed more light into the pathophysiology of CMV infection in patients with CAD in relation to GDF-15 and NrF2 and their implications on disease progression. Ultimately, this would then enable us to identify patients at risk and develop novel strategies for future treatment and prevention of heart diseases in our country. In light of our project research, the question arises whether telomere length could represent a marker of chronic CMV reactivation and uncertainty their length will be modified by the effect of DPP-4 or not?

DETAILED DESCRIPTION:
1. We are aiming to establish a marker for chronic reactivation and pathophysiology of CMV infection in patients with coronary artery disease.
2. We will be able to answer whether there is a link between the seropositive CMV, telomere length, and CAD.
3. We will correlate the seropositive CMV with telomere length, GDF-15 & NRF2.
4. We will detect the origin of our biomarkers by human umbilical vein endothelial cells(HUVECS).
5. We will measure the effect of DPP4-I (on TL & GDF-15 on cardiac cell line).
6. We are looking to establish a new potential risk marker from our study, (GDF-15 & NRF2) which could be tested in a larger cohort of patients. This would then enable us to identify CMV-seropositive patients at risk and develop novel strategies for future treatment and prevention.

ELIGIBILITY:
Inclusion Criteria:

1. According to American Heart Association, patients with a manifestation of myocardial ischemia and angina or angina equivalent (chest pain, abnormal stress testing) with or without T2DM.
2. All patients with risk factors such as hypertension, hyperlipidemia and smokers.

Exclusion Criteria:

1. Psycological disorders
2. Cancers.
3. Strock.
4. Acute and chronic inflammation and Autoimmune diseases were excluded from the study.

Ages: 25 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: The patients will be selected from Cardiology Department in Assiut University Hospital, according to American Heart Association, patients with manifestation of myocardial ischemia and angina or angina equivalent (chest pain, abnormal stress testing) with or without T2DM. All patients with risk factors such as hypertension, hyperlipidemia and smokers.
  The sample size was calculated using EPi Info 2000, version 1.1.2 (Center for disease control and prevention, Atlanta, Georgia, USA) based on proportion of telomere shortening in normal subjects range from 0-1% and it is expected to be 14 % in patients with coronary artery disease (Daily News, American Heart Association, 2016) using 90% confidence interval and 80% power, the sample size is 54 cases of coronary artery disease and 54 control subjects (total 108).
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-10-15 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
Role of endothelial bio markers in patients with coronary artery disease | two years
  genetic expression of new bio markers in coronary artery diseases

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Qi Nan W, Ling Z, Bing C. The influence of the telomere-telomerase system on diabetes mellitus and its vascular complications. Expert Opin Ther Targets. 2015 Jun;19(6):849-64. doi: 10.1517/14728222.2015.1016500. Epub 2015 Feb 13. PMID 25677239